CLINICAL TRIAL: NCT06191120
Title: FAPI Molecular Imaging for Diagnosis of the CMS4 Unfavorable Colorectal Cancer Subtype
Acronym: FoCus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Marnix G.E.H. Lam, MD, PhD, Prof. Dr., UMC Utrecht
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: U23-0607; 2023-509183-17 (EudraCT Number)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Cancer to Liver
Keywords: CMS4; FAPI; Imaging
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: FoCus is a prospective monocenter, proof-of-concept, observational clinical study with a cross-sectional design to address the primary objective, and a longitudinal part to address secondary and exploratory objectives.
  Participant will receive up to three [18]F-ALF-FAPI-74 PET/CT scans, dependent on standard-of-care procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- One [18F]-ALF-FAPI-74 PET/CT scan (Experimental): For patients presenting with metachronous disease, or synchronous disease without the need for two separate surgical sessions for removal of all lesions (i.e. separate liver and primary cancer surgery), and who do not receive any chemotherapy before surgery, only one pre-surgical [18F]-ALF-FAPI-74 PET/CT will be performed.
  Interventions: Radiation: [18F]-ALF-FAPI-74 PET/CT scan
- Two [18F]-ALF-FAPI-74 PET/CT scans (Experimental): For patients presenting with synchronous disease who require two separate surgical sessions (i.e. separate liver and primary cancer surgery), and who do not receive pre-surgical chemotherapy, an [18F]-ALF-FAPI-74 PET/CT will be performed before each surgical session.
  Interventions: Radiation: [18F]-ALF-FAPI-74 PET/CT scan
- Pre-treated group, two [18F]-ALF-FAPI-74 PET/CT scans (Experimental): For patients presenting with metachronous disease, or synchronous disease without the need for two separate surgical sessions for removal of all lesions (i.e. separate liver and primary cancer surgery), and who receive pre-surgical chemotherapy, two [18F]-ALF-FAPI-74 PET/CTs are performed: one before chemotherapy and one before surgery.
  Interventions: Radiation: [18F]-ALF-FAPI-74 PET/CT scan
- Pre-treated group, three [18F]-ALF-FAPI-74 PET/CT scans (Experimental): For patients presenting with synchronous disease who require two separate surgical sessions (i.e. separate liver and primary cancer surgery), and who do receive pre-surgical chemotherapy, three [18F]-ALF-FAPI-74 PET/CTs will be performed: one before chemotherapy and one before each surgical session.
  Interventions: Radiation: [18F]-ALF-FAPI-74 PET/CT scan

INTERVENTIONS:
Radiation: [18F]-ALF-FAPI-74 PET/CT scan — Participants will receive up to three [18F]-ALF-FAPI-74 PET/CT scans. [18F]-ALF-FAPI-74 is a PET tracer with high binding specificity and selectivity to FAP-expressing cells.

SUMMARY:
Colorectal cancer (CRC) is the 3rd most common cancer worldwide and accounts for ~14,000 new diagnoses and ~5,000 deaths in the Netherlands yearly (1.9 million and 935 thousand on a global level). Large scale transcriptional profiling of primary CRC tumors has revealed the presence of four distinct consensus molecular subtypes (CMSs). The CMS4 subtype is associated with a poor prognosis, especially in early CRC, and may benefit less from several standard systemic treatments (e.g. oxaliplatin, 5-fluorouracil, cetuximab), while being relatively sensitive to irinotecan. This is relevant as in the metastatic setting often the first choice first-line systemic therapy regimen is oxaliplatin and not irinotecan-based. Furthermore, tumor cells can acquire a CMS4 phenotype following exposure to chemotherapy, which may contribute to therapy resistance.

CMS4 accounts for ~25% of all early-stage CRC patients and is more prevalent in advanced disease stages (~40% in stage IV CRC). Currently available CMS4 diagnostic tests require tumor tissue samples. The interpretation of biopsy-based CMS4 diagnosis is however complicated by large intra- and inter-lesion heterogeneity of CMS4 status. Extensive biopsy protocols could address the problem of CMS4 heterogeneity but are challenging in routine clinical practice. The development of CMS4-targeted therapy strategies therefore requires a more robust and clinically applicable diagnostic test for comprehensive quantitative assessment of CMS4 status of all lesions - primary and metastatic - in individual cancer patients.

A promising solution for such a diagnostic test is to use a radiotracer that enables the quantitative assessment of CMS4 in vivo by whole body molecular imaging. This technique is particularly suited to assess biomarkers with heterogeneous expression: for diagnostic purposes, as a companion diagnostic for (targeted) therapies, or as part of a 'theranostic' strategy where patient selection using the diagnostic radiotracer is followed by treatment with the same tracer labeled to a therapeutic compound.

Radiolabeled fibroblast activating protein inhibitor (FAPI) is an emerging diagnostic radiotracer that allows the comprehensive whole-body, whole-tumor assessment of fibroblast activation protein (FAP) expression in humans with a very low background uptake also at frequent CRC metastatic sites including the liver. FAP is an excellent candidate molecular imaging target for CMS4, as it is highly expressed on cancer-associated fibroblasts (CAF) that are abundantly present in this CRC subtype. Indeed, the investigators found that FAP gene-expression measured in tumor biopsies - as a single marker - accurately discriminates CMS4 from other CRC subtypes (area under the receiver operating characteristic curve (AUROC): 0.91; 95% confidence interval (CI): 0.90-0.93). The FoCus study will aim to take a next step by relating in vivo assessed FAP protein-expression by [18F]-ALF-FAPI-74 positron emission tomography (PET) / computed tomography (CT) to CMS4 status in patients eligible for colorectal liver metastatectomy as a first proof of concept. Ultimately this will contribute to the development of a diagnostic tool for the comprehensive assessment of CMS4 load in patients with (metastatic) CRC by using [18F]-ALF-FAPI-74 PET/CT molecular imaging, to guide CMS4 subtype-directed therapy decisions.

DETAILED DESCRIPTION:
CRC is the 3rd most common cancer worldwide and accounts for ~14,000 new diagnoses and ~5,000 deaths in the Netherlands yearly (1.9 million and 935 thousand on a global level). CRC is a heterogeneous disease in terms of prognosis, therapy response, and the underlying tumor biology. Large scale transcriptional profiling of primary CRC tumors has revealed the presence of four distinct consensus molecular subtypes (CMSs), which is currently the most robust molecular classification system for CRC. This classification system shows important associations with clinical variables such as primary tumor location, histopathological grade, and prognosis. CMS4 accounts for ~25% of all early-staged CRC patients and is more prevalent in advanced disease stages (~40% in stage IV). Moreover, the CMS4 subtype is characterized by a poor prognosis (e.g. relapse-free survival hazard ratio (HR) of ~1.75 compared to the other subtypes), especially in early CRC, and may benefit less from (often oxaliplatin based) standard systemic treatment regimens. Interestingly, CMS4 CRC seems to benefit more from irinotecan-based chemotherapy regimens. This is relevant as in the metastatic setting often the first choice first-line systemic therapy regimen is oxaliplatin and not an irinotecan-based regimen. Additionally, tumor cells may acquire a CMS4 phenotype following exposure to (fluoropyrimidine-based) chemotherapy, which could contribute to therapy resistance. So far, no effective CMS4-targeted therapies are available for clinical use, although this is an active area of research. For instance, it was recently shown in primary colon cancer that imatinib may have value as CMS-switching (CMS4 to CMS2) drug, characterized by gene expression changes associated with improved survival. Moreover, the MoTriColor study is investigating a TGF-β receptor inhibitor (galunisertib) in combination with capecitabine in patients with advanced chemotherapy resistant CRC with an activated transforming growth factor beta (TGF-β) signature, which is typically activated in the CMS4 CRC subtype (NCT04031872). Finally, as mentioned before, CRC patients with a high CMS4 load could benefit more from an irinotecan-based compared to an oxaliplatin-based treatment regimen.

The genetic signatures upregulated in CMS4 tumors are genes related to TGF-β signaling, epithelial to mesenchymal transition and stromal invasion to which CAFs contribute. In the past decade the effect of the tumor stroma on tumor biology has been studied extensively. The most prominent cell in tumor stroma is the CAF. One of the cell surface markers that distinguish CAFs from normal fibroblasts is FAP.

FAP is expressed during embryogenesis and wound healing. On healthy adult tissues there is almost no expression of FAP. However, FAP is overexpressed on CAFs in the tumor stroma of many different solid tumors. It enables tumor cell migration through extracellular matrix remodeling and has been described to be pro-angiogenic and immunosuppressive in the tumor microenvironment. High FAP expression is associated with a worse overall survival in many epithelial cancers, including CRC. High FAP expression based on IHC of primary CRC tumor samples is associated with poor survival (HR: 1.72, 95% CI: 1.58-9.48, p = 0.009).

In 2018, the first clinical data of a new radiotracer targeting FAP was published. This radiotracer, [68Ga]-FAPI, is based on a quinoline small molecule FAP inhibitor: FAPI. In the last five years, FAPI imaging data of over 3000 cancer patients with many different cancer types were published. Also, multiple publications reported on FAP-targeted radioligands used as last resort therapy with Yttrium-90, Lutetium-177 ([177Lu]) or Samarium-153, with some patients showing stable disease for several months. A first phase I trial investigating [177Lu]-DOTA-FAPI is currently recruiting (NCT04849247). Moreover, another group has recently conducted several first-in-human studies with [177Lu]-radiolabeled FAP inhibitors, further showing the potential of theranostic therapy using FAPI compounds.

Albeit data are still scarce, three studies related tumor FAPI-uptake with FAP-expression by IHC, and all showed a significant positive correlation (r = 0.43-0.94). One study compared this correlation between tissues obtained through resection or biopsy and found the correlation to be stronger following resection. This shows that the sampling method is important due to the heterogeneous expression of FAP within a tumor.

A low background activity and high tumor uptake of FAPI results in exceptionally clear tumor delineation, awarding [68Ga]-FAPI PET with the Society of Nuclear Medicine and Molecular Imaging Image of the Year in 2019. Up to now, [68Ga]-FAPI PET data of 68 patients with (metastatic) CRC was published. Uptake values were high in primary and metastatic CRC, with very low background uptake, including in the normal liver (see also section 4.1b for more information). Furthermore, there is large variation in FAPI uptake in CRC (e.g. SUVmax standard deviation of 3.6 across CRC liver metastases), indicating that variation of FAP-expression can be visualized.

The development of CMS4-targeted therapy strategies for this unfavorable CRC subtype requires a robust and clinically applicable diagnostic test for comprehensive quantitative assessment of CMS4 status of all lesions - primary and metastatic - in individual cancer patients. A 273-gene classifier based on RNA-sequencing of tumor biopsies is the current reference standard to diagnose CMS4, but alternative tests have been developed. All these tests require tumor samples and interpretation is complicated due to intra- and inter-lesion heterogeneity of CMS status. For example, using one of these tests, a study performed by our group found that 55% of 20 studied primary CRC tumors showed both CMS4 positive and negative tumor regions, and CMS4 status can differ substantially between primary and metastatic tumor sites within the same patient. Furthermore, this study showed that multi-region tumor biopsies during colonoscopy to prospectively select CMS4 CRC patients to study the potential of imatinib as a CMS4-specific treatment in a pre-operative proof-of-concept window study confirmed - again - extensive intra-tumor CMS4 heterogeneity.

Beyond this spatial CMS4 heterogeneity, CMS4 may also show temporal heterogeneity during chemotherapy as another study performed by our group has shown in 129 primary CRCs and paired liver metastases, where neoadjuvant chemotherapy was an independent risk factor for the CMS4 subtype. An observation that was corroborated by experimental work on patient-derived CRC organoids: exposure of such organoids to six short cycles of 5-fluorouracil in vitro induced a mesenchymal-like (CMS4) gene-signature. This signature was related to poor prognosis in a large set of CRC patients with publicly available gene-expression data.

Extensive tissue biopsy protocols could address this problem of CMS heterogeneity to allow accurate CMS4 diagnosis but are challenging in routine clinical practice and burdensome for patients. A promising alternative for a CMS4 diagnostic test would be to use a radiotracer that enables the quantitative assessment of CMS4 in vivo by whole body molecular imaging. This imaging modality is particularly suited to assess biomarkers with heterogeneous expression: for diagnostic purposes, as a companion diagnostic for (targeted) therapies, or as part of a 'theranostic' strategy where patient selection using the diagnostic radiotracer is followed by treatment with the same tracer labeled to a therapeutic compound. FAP is an excellent candidate molecular imaging target for CMS4, as it is highly expressed on CAFs that are abundantly present in this CRC subtype. Indeed, FAP gene-expression measured in tumor biopsies - as a single marker - accurately discriminated CMS4 from other CRC subtypes (AUROC: 0.91; 95% CI: 0.90-0.93). Furthermore, reanalysis of published data showed marked [68Ga]-FAPI uptake heterogeneity within and between 15 CRC patients and tumor sites, confirming the potential value of this tracer to diagnose CMS4 CRC.

The FoCus study will take the next step by relating in vivo assessed FAP protein-expression by [18F]-ALF-FAPI-74 PET/CT to CMS4 status. The investigators previously have gained experience with [68Ga]-FAPI-46 imaging by clinically introducing it in the Netherlands in April 2021 - as the first group - in collaboration with SOFIE iTheranostics (the global license holder of FAPI tracers). Up till September 2023, 20 cancer patients with a diagnostic dilemma have been imaged, to which the scan contributed meaningful in all. None of the patients experienced any adverse effects, and - as expected from the literature - tumor-to-background ratios were excellent. Fluoride-18 ([18F]) imaging is superior to Gallium-68 ([68Ga]) with respect to image quality, contrast, harmonization and accessibility for routine use. For these reasons, this study will move forwardwith [18F]-ALF-FAPI-74, produced by Cyclotron Noordwest BV in collaboration with SOFIE iTheranostics.

The relation between [18F]-ALF-FAPI-74 PET/CT and tumor lesion-level CMS4 status specifically in patients who are eligible for CRC liver metastatectomy will be studied, as 1) CMS4 is more prevalent in stage IV disease thereby improving statistical efficiency compared to lower CRC stages; 2) patients often have multiple liver metastases, and if synchronous disease also a primary tumor that will be surgically removed, further improving the effective sample size on a lesion-level and also allowing the evaluation of within-patient heterogeneity. This patient population is therefore ideal for a proof-of-concept. However, results regarding the diagnostic value of [18F]-ALF-FAPI-74 PET/CT for lesion-level CMS4 status obtained from this particular CRC patient subgroup may generalize towards and therefore be clinically relevant for other CRC disease stages and manifestations.

If FoCus shows that [18F]-ALF-FAPI-74 PET/CT is indeed a robust diagnostic test to assess CMS4 load in metastatic CRC patients, its subsequent application as integral biomarker for patient selection is envisioned - without the need for extensive tissue sampling - in clinical studies to develop and evaluate CMS4 subtype-targeted treatment strategies for (metastatic) CRC. This includes theranostic strategies where FAPI itself serves as the targeting moiety for therapeutic compounds. These efforts could ultimately lead to improved personalized CMS4-treatment strategies, patient outcome and quality of life of CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Candidates for liver metastatectomy at the time of liver metastasis diagnosis as clinically indicated in the tumor board (RAKU).
* Patients must have given written informed consent.
* At least one liver metastasis should have a longest diameter of a least 1.5 cm as measured on routinely performed imaging (e.g. magnetic resonance imaging, CT-scan or ultrasound). This minimum diameter will guarantee sufficient tissue material for analysis and will prevent underestimation of [18F]-ALF-FAPI-74 uptake due to partial volume effects.
* CRC patients who received prior treatment before clinical indication for surgical liver metastases resection (both synchronous and metachronous patients, as well as a re-resection of liver metastatic disease) are allowed to enter the study. This is because our prime interest is in the relation between FAPI uptake and the presence of CMS4 at the same point in time, which will likely not be biased by earlier therapies.
* It is allowed for patients to receive concurrent radiofrequency ablation or other local treatments directed to other metastatic disease locations, if at least one liver metastasis of sufficient size is planned to be surgically removed and therefore available for tissue analysis.
* It is allowed for patients to be treated with pre-surgical radiotherapy directed to the primary tumor (e.g. in rectal cancer patients).

Exclusion Criteria:

* Pregnancy.
* Patients treated with a pre-surgical chemotherapy regimen that does not include a fluoropyrimidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Tumor-level CMS4 status as assessed by the current RNA-sequencing based CMS4 status reference standard performed on fresh-frozen tissue samples following surgery. | 1-10 months (dependent on standard-of-care)
  To assess the discriminative ability of pre-surgical in vivo [18F]-ALF-FAPI-74 uptake for CMS4 CRC on a tumor lesion-level in patients eligible for colorectal liver meta-statectomy

SECONDARY OUTCOMES:
FAP protein expression per lesion measured by Enzyme-linked Immunosorbent Assay (ELISA) and immunohistochemistry (IHC) | 1-10 months (dependent on standard-of-care)
  To validate [18F]-ALF-FAPI-74 uptake as a measure of actual histopathologic FAP protein expression
The occurrence, type, and severity of (serious) adverse events (none expected) | 1-10 months (dependent on standard-of-care)
  To contribute to safety data regarding the clinical use of [18F]-ALF-FAPI-74
[18F]-ALF-FAPI-74 standardized uptake values in reference liver and blood pool according to different body-composition correction formulas | 1-10 months (dependent on standard-of-care)
  To evaluate the optimal body-composition correction method for [18F]-ALF-FAPI-74 tracer uptake value standardization
Change in the [18F]-ALF-FAPI-74 standardized uptake values per lesion during chemotherapy | 1-10 months (dependent on standard-of-care)
  To study changes in [18F]-ALF-FAPI-74 uptake during chemotherapy
10-120 minutes post-injection dynamic [18F]-ALF-FAPI-74 uptake levels in tumor lesions and reference organs | 1-10 months (dependent on standard-of-care)
  To evaluate the optimal post-tracer-injection [18F]-ALF-FAPI-74 scan time

OTHER OUTCOMES:
[18F]-ALF-FAPI-74 standardized uptake values measured in volumes of interest (VOIs) within targeted and non-targeted tissues | 1-10 months (dependent on standard-of-care)
  To assess the biodistribution of [18F]-ALF-FAPI-74 (targeting as well as non-targeting) and their determinants as a step towards a theranostic strategy
Site-specific recurrence free survival | 5 years
  To explore relations between pre-surgical [18F]-ALF-FAPI-74 uptake and patient outcome
Overall survival | 5 years
  To explore relations between pre-surgical [18F]-ALF-FAPI-74 uptake and patient outcome
Histologic tumor response: Five-tier Mandard tumor regression grade scale | 1-10 months (dependent on standard-of-care)
  To explore whether change in [18F]-ALF-FAPI-74 uptake during chemotherapy is a possible marker of resistance
RECIST v1.1 response assessment | 1-10 months (dependent on standard-of-care)
  To explore whether change in [18F]-ALF-FAPI-74 uptake during chemotherapy is a possible marker of resistance
Expression of CAF subtype markers such as (ACTA2, CXCL8, CXCL1, MMP1, MMP3, CXCL14, BMP4, COL1A1, FN1, GREM1, RSPO3) measured by IHC or RNA in-situ hybridization on tissue samples following surgery | 1-10 months (dependent on standard-of-care)
  To gain insight into the relationship of FAP expression and [18F]-ALF-FAPI-74 uptake with the presence of distinct CAF subtypes
Tumor-stroma ratio according to van Pelt et al. | 1-10 months (dependent on standard-of-care)
  To gain insight into the relationship of FAP expression and [18F]-ALF-FAPI-74 uptake with the presence of distinct CAF subtypes
[18F]-ALF-FAPI-74 standardized uptake values measured in VOIs within targeted and non-targeted tissues | 1-10 months (dependent on standard-of-care)
  To explore relations between [18F]-ALF-FAPI-74 uptake and various clinicopathological and molecular data
RNA-sequencing derived gene-expression levels per tumor lesion | 1-10 months (dependent on standard-of-care)
  To explore differences in gene-expression (signatures) between tumor lesions with high and low [18F]-ALF-FAPI-74 uptake

CONTACTS AND LOCATIONS:
Overall Officials: M. G.E.H. Lam, Principal Investigator — UMC Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guinney J, Dienstmann R, Wang X, de Reynies A, Schlicker A, Soneson C, Marisa L, Roepman P, Nyamundanda G, Angelino P, Bot BM, Morris JS, Simon IM, Gerster S, Fessler E, De Sousa E Melo F, Missiaglia E, Ramay H, Barras D, Homicsko K, Maru D, Manyam GC, Broom B, Boige V, Perez-Villamil B, Laderas T, Salazar R, Gray JW, Hanahan D, Tabernero J, Bernards R, Friend SH, Laurent-Puig P, Medema JP, Sadanandam A, Wessels L, Delorenzi M, Kopetz S, Vermeulen L, Tejpar S. The consensus molecular subtypes of colorectal cancer. Nat Med. 2015 Nov;21(11):1350-6. doi: 10.1038/nm.3967. Epub 2015 Oct 12. PMID 26457759
- [Background] Trumpi K, Ubink I, Trinh A, Djafarihamedani M, Jongen JM, Govaert KM, Elias SG, van Hooff SR, Medema JP, Lacle MM, Vermeulen L, Borel Rinkes IHM, Kranenburg O. Neoadjuvant chemotherapy affects molecular classification of colorectal tumors. Oncogenesis. 2017 Jul 10;6(7):e357. doi: 10.1038/oncsis.2017.48. PMID 28692036
- [Background] Peters NA, Constantinides A, Ubink I, van Kuik J, Bloemendal HJ, van Dodewaard JM, Brink MA, Schwartz TP, Lolkema MPJK, Lacle MM, Moons LM, Geesing J, van Grevenstein WMU, Roodhart JML, Koopman M, Elias SG, Borel Rinkes IHM, Kranenburg O. Consensus molecular subtype 4 (CMS4)-targeted therapy in primary colon cancer: A proof-of-concept study. Front Oncol. 2022 Sep 6;12:969855. doi: 10.3389/fonc.2022.969855. eCollection 2022. PMID 36147916
- [Background] Lindner T, Loktev A, Altmann A, Giesel F, Kratochwil C, Debus J, Jager D, Mier W, Haberkorn U. Development of Quinoline-Based Theranostic Ligands for the Targeting of Fibroblast Activation Protein. J Nucl Med. 2018 Sep;59(9):1415-1422. doi: 10.2967/jnumed.118.210443. Epub 2018 Apr 6. PMID 29626119
- [Background] Loktev A, Lindner T, Mier W, Debus J, Altmann A, Jager D, Giesel F, Kratochwil C, Barthe P, Roumestand C, Haberkorn U. A Tumor-Imaging Method Targeting Cancer-Associated Fibroblasts. J Nucl Med. 2018 Sep;59(9):1423-1429. doi: 10.2967/jnumed.118.210435. Epub 2018 Apr 6. PMID 29626120
- [Background] Giesel FL, Adeberg S, Syed M, Lindner T, Jimenez-Franco LD, Mavriopoulou E, Staudinger F, Tonndorf-Martini E, Regnery S, Rieken S, El Shafie R, Rohrich M, Flechsig P, Kluge A, Altmann A, Debus J, Haberkorn U, Kratochwil C. FAPI-74 PET/CT Using Either 18F-AlF or Cold-Kit 68Ga Labeling: Biodistribution, Radiation Dosimetry, and Tumor Delineation in Lung Cancer Patients. J Nucl Med. 2021 Feb;62(2):201-207. doi: 10.2967/jnumed.120.245084. Epub 2020 Jun 26. PMID 32591493
- [Background] Lindner T, Altmann A, Giesel F, Kratochwil C, Kleist C, Kramer S, Mier W, Cardinale J, Kauczor HU, Jager D, Debus J, Haberkorn U. 18F-labeled tracers targeting fibroblast activation protein. EJNMMI Radiopharm Chem. 2021 Aug 21;6(1):26. doi: 10.1186/s41181-021-00144-x. PMID 34417894
- [Background] Ubink I, Elias SG, Moelans CB, Lacle MM, van Grevenstein WMU, van Diest PJ, Borel Rinkes IHM, Kranenburg O. A Novel Diagnostic Tool for Selecting Patients With Mesenchymal-Type Colon Cancer Reveals Intratumor Subtype Heterogeneity. J Natl Cancer Inst. 2017 Aug 1;109(8). doi: 10.1093/jnci/djw303. PMID 28376187
- [Background] Strating E, Wassenaar E, Verhagen M, Rauwerdink P, van Schelven S, de Hingh I, Rinkes IB, Boerma D, Witkamp A, Lacle M, Fodde R, Volckmann R, Koster J, Stedingk K, Giesel F, de Roos R, Poot A, Bol G, Lam M, Elias S, Kranenburg O. Fibroblast activation protein identifies Consensus Molecular Subtype 4 in colorectal cancer and allows its detection by 68Ga-FAPI-PET imaging. Br J Cancer. 2022 Jul;127(1):145-155. doi: 10.1038/s41416-022-01748-z. Epub 2022 Mar 16. PMID 35296803
- [Background] Mori Y, Haberkorn U, Giesel FL. 68Ga- or 18F-FAPI PET/CT-what it can and cannot. Eur Radiol. 2023 Nov;33(11):7877-7878. doi: 10.1007/s00330-023-09715-9. Epub 2023 May 12. No abstract available. PMID 37171487
- [Background] Watabe T, Naka S, Tatsumi M, Kamiya T, Kimura T, Shintani Y, Abe K, Miyake T, Shimazu K, Kobayashi S, Kurokawa Y, Eguchi H, Doki Y, Inohara H, Kato H, Mori Y, Cardinale J, Giesel FL. Initial Evaluation of [18F]FAPI-74 PET for Various Histopathologically Confirmed Cancers and Benign Lesions. J Nucl Med. 2023 Aug;64(8):1225-1231. doi: 10.2967/jnumed.123.265486. Epub 2023 Jun 2. PMID 37268427
- [Background] Loktev A, Lindner T, Burger EM, Altmann A, Giesel F, Kratochwil C, Debus J, Marme F, Jager D, Mier W, Haberkorn U. Development of Fibroblast Activation Protein-Targeted Radiotracers with Improved Tumor Retention. J Nucl Med. 2019 Oct;60(10):1421-1429. doi: 10.2967/jnumed.118.224469. Epub 2019 Mar 8. PMID 30850501